CLINICAL TRIAL: NCT05536908
Title: Evaluating the Impact of Supplementing Residential Substance Use Treatment With Written Exposure Therapy for Veterans With Co-Occurring PTSD and Substance Use Disorders
Brief Title: Evaluating Supplementing Residential Substance Use Treatment With Written Exposure Therapy for Veterans With Post Traumatic Stress Disorder (PTSD) and Substance Use Disorders (SUD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Boston Healthcare System (U.S. Federal Agency); Center for Biostatistics and Health Data Science (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D4083-P; I21RX004083-01A1 (NIH)
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: PTSD; Substance Use Disorders
Keywords: PTSD; Substance Use Disorders; Treatment; Comorbidity
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: 50 Veterans are assigned to the combined PTSD/ residential substance use treatment (resWET) or Treatment as Usual (TAU: residential substance use treatment program). Two small sub-studies were approved as followup studies: 1) to recruit participants from the larger study to evaluate them over a long-term followup period (up to 20 of the original participants). 2) to recruit approximately 10 new participants, 5 who would be randomized to receive the CAPS twice and 5 to have filler measures (WhoDAS and TLFB). All participants will be administered the PHQ-9 and PCL at 4 time points (3 while in the DOM SUD program, and 1 one month following).
Who Masked: Outcomes Assessor
Masking Description: Provider conducting CAPS-5 will not have access to treatment condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- resWET (Experimental): Residential Written Exposure Therapy (resWET): Treatment as Usual (TAU) plus 5-individual Written Exposure Therapy (WET) sessions (40-60 min each; Marx & Sloan, 2019) twice a week for two weeks and once a week for the final session, administered by WET trained psychologists, social workers, or postdoctoral residents. Treatment instructions are read, patients write for 30 minutes, and the writing is briefly processed. No formal written homework is required.
  Interventions: Behavioral: Residential Written Exposure Therapy
- Treatment as Usual (TAU) (Active Comparator): Treatment as Usual (DOM SUD): The DOM SUD (TAU) is a 24-bed intensive substance use disorder (SUD) residential program with a typical 28-day length of stay. The program focuses on evidence-based treatments for SUD such as Cognitive-Behavioral Therapy, Motivational Enhancement Therapy, Medication Assisted Treatment, and Contingency Management therapy. Patients diagnosed with Post-traumatic Stress Disorder (PTSD) are typically referred to outpatient PTSD treatment following DOM SUD and often attend Seeking Safety during the program. Most of the programming is group-based though Veterans also have weekly individual case management appointments.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Residential Written Exposure Therapy — Residential Written Exposure Therapy (resWET): TAU plus 5-individual WET sessions (40-60 min each; Marx & Sloan, 2019) twice a week for two weeks and once a week for the final session, administered by WET trained psychologists, social workers, or postdoctoral residents. Treatment instructions are read, patients write for 30 minutes, and the writing is briefly processed. No formal written homework is required.
  Other Names: resWET
  Arms: resWET
Behavioral: Treatment as Usual — Treatment as Usual (DOM SUD): The DOM SUD (TAU) is a 24-bed intensive SUD residential program with a typical 28-day length of stay. The program focuses on evidence-based treatments for SUD such as Cognitive-Behavioral Therapy, Motivational Enhancement Therapy, Medication Assisted Treatment, and Contingency Management therapy. Patients diagnosed with PTSD are typically referred to outpatient PTSD treatment following DOM SUD and often attend Seeking Safety during the program. Most of the programming is group-based though Veterans also have weekly individual case management appointments.
  Other Names: TAU
  Arms: Treatment as Usual (TAU)

SUMMARY:
Posttraumatic Stress Disorder (PTSD) and Substance Use Disorder (SUD) are highly comorbid, and comorbidity increases risk for poor functional outcomes. Risks for poor quality of life and suicide increase further for those with co-occurring PTSD and SUD diagnoses as compared to either condition alone, with suicide attempt rates three times higher for Veterans with alcohol use disorder and PTSD (Norman, Haller, Hamblen, Southwick & Pietrzak, 2018). For patients with PTSD-SUD, there is evidence of greater PTSD symptom severity and poorer SUD treatment outcomes (e.g., Back et al., 2000), as well as higher rates of homelessness and disability (Bowe & Rosenheck, 2015). PTSD-SUD treatments have shown promising reductions in PTSD and SUD symptoms (Flanagan, Korte, Killeen & Back,2016). Yet, there are still major challenges in widely implementing concurrent or single-target gold-standard treatments for this population, especially with rural veterans where care access may be limited (e.g., Flanagan et al., 2016). Written Exposure Therapy (WET) is a front-line, brief and effective treatment for PTSD that addresses some of the challenges posed by other gold-standard treatments. This project is designed to examine the feasibility and acceptability of Written Exposure Therapy (WET) delivered to Veterans with comorbid PTSD-SUD while they are completing a 28 day-residential SUD program (DOM SUD). The preliminary effects of the treatment during the program, and at one month and 3-month follow-up periods will also be examined, with particular attention to rates of substance use, homelessness, treatment attendance, treatment completion, quality of life, suicidality, and PTSD and depression symptoms. Veterans enrolled in the residential substance use disorder clinic will be recruited for screening into the study. Those that meet criteria for PTSD will be randomized into one of two treatment arms: Treatment as Usual (TAU: DOM SUD) and Written Exposure Therapy in a residential SUD program (resWET). Those in the TAU control group will participate in the DOM SUD treatment program, while those in the resWET group will also have five individual treatment sessions of WET. Participants will complete weekly measures of symptoms, in addition to rating cravings for substance use. Treatment completion rates will also be compiled for both DOM SUD and resWET. Participants will complete pre-treatment, post-treatment, 1 month, and 3 month follow-up measures to look for important trends regarding symptom responses to treatment (e.g., PTSD, depression), as well as suicide attempts, homelessness, treatment attendance, treatment completion, substance use, and quality of life. This preliminary data will be used to inform future studies. Additionally, providers will provide feedback to provide essential information about implementation barriers that need to be addressed for the broader uptake of the treatment approach and to enhance accessibility of the treatment. All Veterans will also provide feedback about their treatment. Findings will be used to improve the treatment and assessment approach and to prepare for a larger study to evaluate resWET.

DETAILED DESCRIPTION:
Posttraumatic Stress Disorder (PTSD) and Substance Use Disorder (SUD) are highly comorbid, and comorbidity increases risk for poor functional outcomes. SUDs are associated with poor functional outcomes, such as quality of life, community engagement, and suicide (Teeters, Lancaster, Brown & Back, 2017). Risks for poor quality of life and suicide increase further for those with co-occurring PTSD and SUD diagnoses as compared to either condition alone, with suicide attempt rates three times higher for Veterans with alcohol use disorder and PTSD (Norman, Haller, Hamblen, Southwick & Pietrzak, 2018). For patients with PTSD-SUD, there is evidence of greater PTSD symptom severity and poorer SUD treatment outcomes (e.g., Back et al., 2000), as well as higher rates of homelessness and disability (Bowe & Rosenheck, 2015). PTSD-SUD treatments have shown promising reductions in PTSD and SUD symptoms (Flanagan, Korte, Killeen & Back, 2016). Yet, there are still major challenges in widely implementing concurrent or single-target gold-standard treatments for this population, especially with rural veterans where care access may be limited (e.g., Flanagan et al., 2016). Written Exposure Therapy (WET) is a front-line, brief and effective treatment for PTSD that addresses some of the challenges posed by other gold-standard treatments. This project is designed to examine the feasibility and acceptability of Written Exposure Therapy (WET) delivered to Veterans with comorbid PTSD-SUD while they are completing a 28 day-residential SUD program (DOM SUD). The preliminary effects of the treatment during the program, and at one month and 3-month follow-up periods will also be examined, with particular attention to rates of substance use, homelessness, treatment attendance, treatment completion, quality of life, suicidality, and PTSD and depression symptoms. Veterans enrolled in the DOM SUD with PTSD Checklist-5 (PCL-5) scores over 33 will be recruited for further screening into the study. Those that meet criteria for PTSD through confirmation using the Clinician Administered PTSD Scale for DSM-5 (CAPS-5) will be randomized into one of two treatment arms: Treatment as Usual (TAU: DOM SUD) and Written Exposure Therapy in a residential SUD program (resWET). Randomization will be stratified by gender and oversampling for women and minority participants will be used. Those in the TAU control group will participate in the DOM SUD treatment program, while those in the resWET group will also have five individual treatment sessions of WET. Participants will complete weekly measures of symptoms, in addition to rating cravings for substance use. Treatment completion rates will also be compiled for both DOM SUD and resWET. Participants will complete pre-treatment, post-treatment, 1 month, and 3 month follow-up measures in person, over video, or by phone, and these measures, along with data available from the treatment record, will be examined using descriptive analyses to look for important trends regarding both symptom responses (e.g., PTSD, depression) to treatment, as well as behavioral and functional outcomes (such as suicide attempts, homelessness, treatment attendance, treatment completion, substance use, quality of life). This preliminary data will be used to inform future studies using this treatment approach. Additionally, providers in the DOM SUD will complete treatment feasibility and satisfaction surveys and focus groups to provide essential information about implementation barriers that need to be addressed for the uptake of the treatment approach and to enhance the accessibility of the treatment. All Veterans will also provide feedback about their treatment, through survey when the treatment is complete, and focus group participation. Findings from both qualitative and quantitative data will be used to improve the treatment and assessment approach and to determine effect sizes of key measures (World Health Organization- Disability Assessment Schedule (WHO-DAS), PTSD Checklist (PCL), Patient Health Questionnaire (PHQ-9)) to prepare for a fully powered randomized control trial (RCT) to systematically evaluate resWET.

Two small sub-studies were approved and added: 1) as a longer term follow-up, study staff reached out to prior participants to re-evaluate their symptoms using the same measures. Participants were reconsented for this additional time period as it was not a part of the original study. 2) A small group of Veterans enrolled in the residential substance use treatment program were recruited for a follow-up study to evaluate the impact of administering a clinician interview for PTSD on PTSD and depressive symptoms at four time points.

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses of a substance use disorder (SUD) and PTSD
* Enrolled in the residential substance use disorder treatment program (DOM SUD) at the Salem VAMC

Exclusion Criteria:

* Current Manic Episode
* Current Suicidal Intent
* Previous Written Exposure treatment
* Unable to write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2026-01-05 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | Week 4
  Standardized patient treatment satisfaction measure, used in substance use treatment settings (Kelly et al, 2018). 8 items measuring satisfaction with treatment, Likert scales from 1 (low satisfaction) to 4 (high satisfaction). Total scores range from 8 to 32, with higher scores indicating greater satisfaction. High concurrent validity and internal consistency. Average item scores of 3 or higher indicate satisfaction with treatment. Completed by participants at the conclusion of 28 day program.
Acceptability of Intervention Measure (AIM) | Week 4
  Four item Likert scale, ranging from 1-5, with higher scores indicating greater acceptability of intervention. Completed by program staff and WET providers at the conclusion of treatment. Average scores of 4 or higher on each measure will be used as our criterion for acceptability.
Change in World Health Organization-Disability Assessment Schedule (WHO-DAS 2.0) | Week 1, 4, 8, 16
  A 36-item self-report measure of functioning in several areas: Understanding and Communicating, Getting Around, Self-Care, Getting Along with People, Life Activities, and Participation in Society. This measure has high internal consistency, high test-retest reliability, and good concurrent validity. Items are rated on a 5-point Likert scale ranging from 0-4. Higher scores are indicative of greater functional disability. 0 score indicates no disability and 100 means full disability. Subscales include: Cognition, Mobility, Self-care, Getting Along, Life Activities (household), Life Activities (work/school), and Participation. Each subscale has a range from 0 to 100 as above.
Change in PTSD Checklist-5 (PCL-5) | Weeks 1, 2, 3, 4, 8, 16
  20-item self-report measure that assesses for DSM-5 symptoms of PTSD. Items are responded to on a 5-point Likert scale ranging from 0-4. Total scores range from 0-80 with higher scores indicative of greater symptom severity. A cut-off score of 33 is often used to determine clinical significance of symptoms . The scale has strong internal consistency, good convergent validity, and acceptable discriminant validity. It is also sensitive to change and can be used to track treatment related changes over time.
Change in Clinician Administered PTSD Scale for DSM-5 (CAPS-5) | Week 1, 4, 8, 16
  A gold-standard 30-item clinician administered structured interview used to make diagnoses of PTSD. Severity score based on 20 items, ranging from 0-4, with higher scores indicating greater severity. Range from 0-80.
Change in Patient Health Questionnaire-9 (PHQ-9) | Weeks 1, 2, 3, 4, 8, 16
  A 9 item self-report measure of depressive symptoms, with a 10th item assessing symptom associated distress. Items are rated on a 4-point Likert scale ranging from 0-3. Scores range from 0-30 with higher scores indicative of greater symptom severity. This measure is shown to have high internal validity and strong predictive validity. Cut off scores greater or equal to 10 are used to determine clinical significance of symptoms.
Change in Brief Addition Monitor (BAM) | Week 1, 4, 8, 16
  A 17-item self-report measure that provides scores on three factors: Recovery Protection, Physical and Psychological Problems, and Substance Use and Risk. Each shown to be responsive to treatment related change. The measure shows acceptable psychometric properties. Items are scored from 0 to 4, with a range from 0 to 68. Higher scores are indicative of more difficulties.
Change in Timeline Follow Back for Substance Use (TLFB) | Weeks 1, 4, 8, 16
  A calendar-based follow-back method to provide continuous measure of substance use. This detailed procedure elicits daily information on substance use and has been found reliable. The main outcome measures will be percentage of participants abstinent for each follow-up period and mean number of days abstinent. A tally of days using alcohol, drugs, and polysubstance use are computed, with a range of 0 for no days used over 30 day period, to 30 with daily use.
Treatment Attendance | Week 16
  Treatment attendance (number of WET sessions attended out of those scheduled vs. case management sessions attended vs. scheduled). Converted to percentage (sessions attended/ scheduled). Higher numbers indicate better attendance, range from 0-100.
Intervention Appropriateness Measure (IAM) | Week 4
  4 item Likert scale, ranging from 1-5, with higher scores indicating greater appropriateness. Completed by program staff and WET providers at the conclusion of treatment. Average scores of 4 or higher on each measure will be used as our criterion for appropriateness.
Feasibility of Intervention Measure (FIM) | Week 4
  4 item Likert scales, ranging from 1-5, with higher scores indicating greater intervention feasibility. Completed by program staff and WET providers at the conclusion of treatment. Average scores of 4 or higher on each measure will be used as our criterion for feasibility.
Treatment Completion rates | 4 weeks
  Participants will be categorized into Treatment Completer for WET if all 5 sessions are completed and DOM SUD Treatment Completer if the 28-day program is completed.

SECONDARY OUTCOMES:
Change in Cravings | Weeks 1, 2, 3, and 4
  5 point Likert scale developed for this study. Item ranges from 1 (no craving) to 5 (extreme craving).
Suicide Attempts | Week 16
  Count of suicide attempt(s) denoted by Suicide Behavior Reports from study enrollment through 3 month follow-up.
Homelessness Status | Week 16
  Record review to determine housing status based on CPRS notes and diagnosis special category.
Drug Screen status | Week 16
  Drug screen results through 3 month follow-up period will be captured via record review in CPRS.

OTHER OUTCOMES:
Columbia Suicide Severity Rating Scale | Week 1, 4, 8, and 16
  Used for suicide risk assessment. Includes questions on suicidal ideation, intensity of ideation, and suicidal behavior. The C-SSRS showed strong concurrent validity with documented suicide attempts and showed good predictive validity in predicting future attempts. Used for study eligibility and safety monitoring, no total score or range of score is utilized.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Holohan, Principal Investigator — Salem VA Medical Center, Salem, VA
Locations (1):
- Salem VA Medical Center, Salem, VA, Salem, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data that underlie the results reported in the article.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 9 months and ending after 3 years of article publication.
Access Criteria: Proposals should be directed to: dana.holohan@va,gov. To gain access, data requestors will need to sign a data access agreement and Salem IRB needs to approve the request.

DOCUMENTS (1):
  • Informed Consent Form (2023-09-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT05536908/ICF_000.pdf